CLINICAL TRIAL: NCT03187613
Title: Correlation of Metamorphopsia and Aniseikonia to Retinal Shift Following Retinal Detachment Surgery
Status: Completed | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017/730 REK
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2020-10

CONDITIONS: Retinal Detachment
Keywords: Retinal shift; Aniseikonia; Metamorphopsia; Autofluorescence
MeSH Terms: conditions — Retinal Detachment; Aniseikonia; Vision Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Individuals operated for rhegmatogenous retinal detachment will be prospectively evaluated for postoperative retinal shift. Fundus autofluorescence will be used to evaluate retinal shift that will be correlated to visual acuity, metamorphopsia, aniseikonia, and stereopsis.

ELIGIBILITY:
Inclusion Criteria:

* Acute rhegmatogenous retinal detachment, fovea detached, able to signe

Exclusion Criteria:

* Secondary retinal detachment like tractional, serous or with ora serrata dialysis, fovea on

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals treated at Stavanger University Hospital
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Retinal shift | 2 years
  Measured on fundus autofluorescence

SECONDARY OUTCOMES:
Visual acuity | 6 and 24 months
  Best Corrected Visual Acuity
Metamorphopsia | 6 and 24 months
  M-Chart
Aniseikonia | 6 and 24 months
  New Aniseikonia Test
Stereopsis | 6 and 24 months
  Titmus Test

CONTACTS AND LOCATIONS:
Overall Officials: Vegard Forsaa, MD, Study Director — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Department of Ophthalmology, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Thomseth VM, Lindtjorn B, Ushakova A, Forsaa VA. LONG-TERM CHANGES IN VISUAL FUNCTION AND EN FACE OPTICAL COHERENCE TOMOGRAPHY FINDINGS IN FOVEA-OFF RETINAL DETACHMENT: A 2-Year Prospective Study. Retina. 2023 Feb 1;43(2):330-337. doi: 10.1097/IAE.0000000000003670. PMID 36695802
- [Derived] Thomseth VM, Ushakova A, Krohn J, Utheim TP, Austeng D, Fossen K, Varhaug P, Malmin A, Skeiseid L, Tharaldsen A, Lindtjorn B, Johannesen H, Juul J, Forsaa VA. STRUCTURAL PATHOLOGY AFTER RETINAL DETACHMENT: Multicolor Confocal Scanning Laser Ophthalmoscopy Versus Color Fundus Photography. Retina. 2021 Sep 1;41(9):1958-1965. doi: 10.1097/IAE.0000000000003113. PMID 33464027
- [Derived] Thomseth VM, Engelsvold DH, Ushakova A, Forsaa VA. EN FACE IMAGING OF OUTER RETINAL PATHOLOGY AFTER RETINAL DETACHMENT. Retina. 2021 Feb 1;41(2):324-330. doi: 10.1097/IAE.0000000000002814. PMID 32282661